CLINICAL TRIAL: NCT06391970
Title: Exploring Long-COVID Impact on Cognition Through Digital Neuropsychological Assessment
Brief Title: Digital Cognition Study During Long-COVID
Acronym: DIGICOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: ViewMind (Industry)
Responsible Party: Principal Investigator, Magali Perquin, Researcher, Luxembourg Institute of Health
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20210613; 16758430 (Other Grant/Funding Number: Fonds National de la Recherche (FNR) Luxembourg); 202208/05 (Other: National Research Ethics Committee (CNER) Luxembourg)
Record Dates: First submitted 2024-04-29; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: COVID-19, Long Haul
Keywords: Cognition, Digital Biomarkers, Validation, Cognitive Reserve
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: DigiCog is a crossover interventional study, involving participants selected both with and without the specific condition of long COVID. The intervention in this study is the use of a new digital device, which is being evaluated in comparison to the gold standard method.
  Each participant receives both interventions in a predetermined sequence. This crossover design enables within-subject comparisons, as each participant acts as their own control. By comparing outcomes within the same participant under different interventions, this design helps to reduce variability and increase the statistical power of the study.
  NB: Although a crossover design may typically imply multiple arms, in this specific study, participants serve as their own controls, resulting in only one arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DigiCog Intervention (Other): Although DigiCog participants receive two interventions (the new digital device and the gold standard method), they are not randomized to different intervention groups. Instead, each participant serves as their own control, receiving both interventions sequentially. Therefore, the study has one arm.
  Interventions: Device: Cognitive screening

INTERVENTIONS:
Device: Cognitive screening — The cognitive abilities of participants will be assessed using two different interventions: the first utilizing the new digital device, and the second employing the gold standard method.

SUMMARY:
The persistence of the COVID-19 disease symptoms, such as extreme fatigue, shortness of breath, cardiovascular complications, depression and anxiety, pain, brain fog, loss of taste/smell, headaches as well as loss of memory has been evoked in many studies. This project aims at approaching the persistent symptomatology on cognition, more than 1 year after the infection.

When we refer to cognition, we refer to everything associated with knowledge, that is, the accumulation of information we have acquired through learning or from our experience. We can define cognitive processes as the processes we use to incorporate new knowledge and make decisions based on it. Through these processes several cognitive functions intervene: perception, attention, memory, reasoning, language, learning, decision-making. All of these cognitive functions work together to integrate knowledge as a whole and create an interpretation of the world around us. Usually neuropsychological tests are used to evaluate cognitive problems, they consist in different exercises sometimes with words, figures to draw, images to remember, movement to repeat, numbers to link together etc.

The DigiCog project here propose

1. to test and validate a very novel device, which uses the eyes movement during tasks to evaluate very quickly the cognitive functioning;
2. to study potential cognitive problems long-term after COVID-19; and
3. to explore how cognition could be preserved.

Finally, this project will also help to bring the innovative device tested to the market, for accurately monitoring people with long COVID.

DETAILED DESCRIPTION:
The Digital Cognition study ("DigiCog") will be conducted within the framework of an already existing robust research project, Predi-COVID (NCT04380987), launched in May 2020 by the Luxembourg Institute of Health (LIH). This cohort study has originally enrolled -and is still ongoing- patients with COVID-19 disease and followed them for over a year in order to approach the potential long-term health effects of the pathology, the "chronic post-COVID syndrome", (https://www.lih.lu/blog/our-news-1/post/a-year-of-predi-covid-407#blog_content) or more frequently referred to as "Long COVID" . If the Predi-COVID study has first been devoted to acute and early symptomatology, it now covers a wide range of medical conditions potentially linked to the persistence of COVID-19 disease, such as extreme fatigue, pain, allergy, renal and cardiovascular complications, stress and anxiety, emotions, memory impairment as well as neurological complications. In this context, the working collaboration between LIH and VIEWMIND Company is a major opportunity to incorporate VIEWMIND's technology in a spin-off project, to additionally screen neurocognitive conditions after COVID-19, improving Long COVID diagnosis. The state-of-the-art VIEWMIND's technology (herein referred to as "VMTech") is indeed a non-invasive and reliable digital tool, using artificial intelligence to deliver accurate results especially on cognitive performance, areas of the brain functioning and high-level motor skills, as well as identifying neurocognitive pathologies (see https://www.viewmind.ai/copy-of-terms-of-service; https://ww2.frost.com/news/press-releases/viewmind-applauded-by-frost-sullivan-for-its-one-of-a-kind-digital-biomarker-technology-for-neurocognitive-disorders). Moreover this cognitive screening will be analyzed according to persistent COVID-19 symptomatology, but also in relationship with the initial severity of SARS-COV-2 infection, and individual features and habits of participants. As a multifactorial approach, the project will test VMTech in a research framework on COVID-19, it will additionally use a complementary cognitive battery of tests as the gold standard.

Hence, this collaborative project fits with the expectations and requirements of the funding joint call Healthtech, addressing the need of gathering evidence of effectiveness "in real-life" of the developed tool. The DigiCog project consortium is adequate to validate the digital biomarker technology, being a balanced public private partnership, based on an on-going powerful cohort study, a long lasting expertise in public and precision health, and an advanced and recognized technology. The project will help to bring VMTech to the market for accurately monitoring people with Long COVID.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have previously participated in the Predi-COVID study (Registration number NCT04380987), or who have experienced COVID-19 at least once before 2022.
* Participants who have signed the informed consent form
* Participants aged between 25 and 65 years old

Exclusion Criteria:

* Psychological or neurological disorders history especially those detected before the COVID-19 disease (e.g. epilepsy, stroke, chronic fatigue) as well as treatment that could interfere with the assessment (e.g., antipsychotics, antidepressants, mood stabilizers, antiepileptics, benzodiazepines)
* Poor eyesight, rendering the use of the digital device impossible
* Inability to speak the proposed languages

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive status assessed with the digital device, of individuals with/without symptoms persisting long-term after COVID-19 disease. | Each assessment and evaluation session lasts approximately 20 minutes and occurs once.
Cognitive status assessed with the gold standard procedure, of individuals with/without symptoms persisting long-term after COVID-19 disease. | Each assessment and evaluation session lasts approximately 1 h and occurs once.

CONTACTS AND LOCATIONS:
Overall Officials: Magali PERQUIN, PhD, Principal Investigator — Luxembourg Institute of Health
Locations (1):
- Luxembourg Institute of Health, LCTR, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: Undecided